CLINICAL TRIAL: NCT05192109
Title: Study 2: Learning New Words From Overhearing in Children With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Emerson College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 280522
Record Dates: First submitted 2022-01-03; First posted 2022-01-14 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Addressed (Experimental): Children participate via video in an interaction with an experimenter who uses the word to be learned.
  Interventions: Behavioral: Addressed Speech
- Overheard (Experimental): Children watch via video while an experimenter uses the word to be learned in an interaction with another experimenter.
  Interventions: Behavioral: Overheard Speech

INTERVENTIONS:
Behavioral: Overheard Speech — New words are introduced with the child as a bystander rather directly taught.
  Arms: Overheard
Behavioral: Addressed Speech — New words are introduced directly to the child by an experimenter.
  Arms: Addressed

SUMMARY:
The goal of this research is to explore abilities to learn word meanings from overheard conversations in children with ASD (and, as a control, typically developing children).

Specific Aim 2 (Experiment 2): Determine whether children with ASD can learn from addressed and overheard teaching via videoconferencing. The investigators will use a similar procedure to Study 1, except that both overheard and directed teaching will take place on video.

ELIGIBILITY:
Inclusion Criteria:

children with or without a diagnosis of ASD between 18 to 71 months of age

Exclusion Criteria:

native language is not English born premature (< 36 weeks) has uncorrected hearing or vision impairments has developmental disorders or medical conditions other than ASD that affect language or cognition (excepting psychiatric conditions often comorbid with ASD such as ADHD) has a history of photosensitive epileptic seizures

Ages: 18 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 342 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Emerson College, Boston, Massachusetts
  - New York University, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ASD - Addressed First, Then Overheard: Children with ASD are exposed to new words. Addressed Speech: New words are introduced directly to the child by an experimenter.
  Overheard Speech: New words are introduced while children observe.
- ASD - Overheard First, Then Addressed: Children with ASD are exposed to new words. Overheard Speech: New words are introduced while children observe. Addressed Speech: New words are introduced directly to the child by an experimenter.
- TD - Addressed First, Then Overheard: Children with TD are exposed to new words. Addressed Speech: New words are introduced directly to the child by an experimenter.
  Overheard Speech: New words are introduced while children observe.
- TD - Overheard First, Then Addressed: Children with TD are exposed to new words. Overheard Speech: New words are introduced while children observe. Addressed Speech: New words are introduced directly to the child by an experimenter.
Period: First Behavioral Task (3 Minutes)
Arm/Group | ASD - Addressed First, Then Overheard | ASD - Overheard First, Then Addressed | TD - Addressed First, Then Overheard | TD - Overheard First, Then Addressed
Started | 87 | 89 | 85 | 81
Completed | 78 | 78 | 83 | 79
Not Completed | 9 | 11 | 2 | 2
Not completed — Withdrawal by Subject | 9 | 11 | 2 | 2
Period: Second Behavioral Task (3 Minutes)
Arm/Group | ASD - Addressed First, Then Overheard | ASD - Overheard First, Then Addressed | TD - Addressed First, Then Overheard | TD - Overheard First, Then Addressed
Started | 87 | 89 | 85 | 81
Completed | 78 | 78 | 83 | 79
Not Completed | 9 | 11 | 2 | 2
Not completed — Withdrawal by Subject | 9 | 11 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASD - Addressed First, Then Overheard | ASD - Overheard First, Then Addressed | TD - Addressed First, Then Overheard | TD - Overheard First, Then Addressed | Total
Number analyzed (Participants) | 87 | 89 | 85 | 81 | 342
Age, Continuous [Mean (Standard Deviation); unit: months] | 51.8 (10.6) | 52.1 (10.2) | 41.5 (14.2) | 31.0 (8.2) | 41.7 (14.3)
Sex/Gender, Customized [Number; unit: participants]
  Number of Enrolled Males | 66 | 66 | 47 | 56 | 235
  Number of Enrolled Females | 21 | 22 | 38 | 25 | 106
  Number Prefer not to Answer | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian / Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 4 | 5 | 4 | 3 | 16
  Black | 10 | 5 | 6 | 4 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  White | 42 | 57 | 52 | 56 | 207
  More than one | 16 | 5 | 17 | 14 | 52
  Unknown | 8 | 14 | 2 | 2 | 26
  Hispanic/Latine | 7 | 3 | 2 | 2 | 14
Region of Enrollment [Number; unit: participants]
  United States | 87 | 89 | 85 | 81 | 342

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Time During Which Children's Eye Gaze is Directed Toward the Target Object
Description: Children's eye gaze is recorded as they look at images. The proportion of time during which gaze is directed to an image of the targeted word is the dependent measure.
Time Frame: immediately after viewing 3-minute interaction
Population: Not all enrolled participants were analyzed because of exclusions due to, e.g., experimenter error or children paying insufficient attention.
Measure: Mean (Standard Deviation); unit: proportion of time
Groups:
- ASD - Addressed: Children with ASD are exposed to new words. Addressed Speech: New words are introduced directly to the child by an experimenter.
- ASD - Overheard: Children with ASD are exposed to new words. Overheard Speech: New words are introduced while children observe.
- TD - Addressed: Children with TD are exposed to new words. Addressed Speech: New words are introduced directly to the child by an experimenter.
- TD - Overheard: Children with TD are exposed to new words. Overheard Speech: New words are introduced while children observe.
Arm/Group | ASD - Addressed | ASD - Overheard | TD - Addressed | TD - Overheard
Number analyzed (Participants) | 80 | 82 | 106 | 104
proportion of time | 0.42 (0.35) | 0.44 (0.33) | 0.49 (0.34) | 0.38 (0.31)
Statistical Analysis 1: Comparison: ASD - Addressed vs ASD - Overheard vs TD - Addressed vs TD - Overheard; The primary statistical analysis involves asking whether children's preference to look at the target is significantly greater in one condition and/or group than the other. Mixed-effects regression analyses are used with the proportion-empirical-logit transformed-of target looking as the dependent measure, participant as random effect, and condition and group and their interaction as fixed effects; Test type: Other; p < 0.01, Regression, Linear — This is the p-value for the simple effect of condition
Statistical Analysis 2: Comparison: ASD - Addressed vs ASD - Overheard vs TD - Addressed vs TD - Overheard; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.93, Regression, Linear — This is the p-value for the simple effect of diagnostic group
Statistical Analysis 3: Comparison: ASD - Addressed vs ASD - Overheard vs TD - Addressed vs TD - Overheard; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.01, Regression, Linear — This is the p-value for the interaction between condition and group

2. Primary Outcome: Proportion of Time During Which Children's Eye Gaze is Directed Toward the Target Object
Description: as for outcome 1
Time Frame: 5 minutes after viewing interaction
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of time
Groups:
- ASD - Addressed; TD - Addressed: Children participate in an interaction with an experimenter who uses the word to be learned.
  Addressed Speech: New words are introduced directly to the child by an experimenter.
- ASD - Overheard; TD - Overheard: Children observe while an experimenter uses the word to be learned in an interaction with another experimenter.
  Overheard Speech: New words are introduced with the child as an observer rather directly taught.
Arm/Group | ASD - Addressed | ASD - Overheard | TD - Addressed | TD - Overheard
Number analyzed (Participants) | 73 | 77 | 98 | 92
proportion of time | 0.43 (0.34) | 0.30 (0.32) | 0.42 (0.34) | 0.43 (0.32)
Statistical Analysis 1: Comparison: ASD - Addressed vs ASD - Overheard vs TD - Addressed vs TD - Overheard; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.01, Regression, Linear — This is the p-value for the simple effect of condition
Statistical Analysis 2: Comparison: ASD - Addressed vs ASD - Overheard vs TD - Addressed vs TD - Overheard; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.22, Regression, Linear — This is the p-value for the simple effect of group
Statistical Analysis 3: Comparison: ASD - Addressed vs ASD - Overheard vs TD - Addressed vs TD - Overheard; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.01, Regression, Linear — This is the p-value for the interaction between condition and group

ADVERSE EVENTS:
Time Frame: the duration of study participation (approximately 10 minutes)
Description: Our experimental paradigm involves presenting children with videos of everyday child-friendly actions during a 10-minute interaction. There is no risk of Serious Adverse Events or All-Cause Mortality during the session.
Arm/Group | ASD - Addressed | ASD - Overheard | TD - Addressed | TD - Overheard
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/176 | 0/166 | 0/166
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/176 | 0/166 | 0/166
Other Adverse Events (participants affected / at risk) | 0/176 | 0/176 | 0/166 | 0/166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT05192109/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT05192109/ICF_000.pdf